CLINICAL TRIAL: NCT05076617
Title: An Open-Label, Multicenter, Outpatient Extension Study to Evaluate the Safety and Tolerability of Staccato Alprazolam in Study Participants 12 Years of Age and Older With Stereotypical Prolonged Seizures
Brief Title: A Study to Test the Safety and Tolerability of Staccato Alprazolam in Study Participants 12 Years of Age and Older With Stereotypical Prolonged Seizures
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0165; 2021-002637-42 (EudraCT Number); 2023-508868-30 (Registry Identifier: EU Clinical Trials); U1111-1299-3027 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stereotypical Prolonged Seizures
Keywords: Stereotypical prolonged seizures; Phase 3; Staccato alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Staccato alprazolam (Experimental): Participants will receive Staccato alprazolam by inhalation.
  Interventions: Drug: Staccato alprazolam

INTERVENTIONS:
Drug: Staccato alprazolam — * Pharmaceutical form: Inhalation powder
  * Route of administration: Inhalation
  Participants will receive Staccato alprazolam during the Treatment Period.
  Other Names: UCB7538

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability of Staccato alprazolam.

ELIGIBILITY:
Inclusion criteria:

* Participant must be ≥12 years of age at the time of signing informed consent
* Participant must have a study caregiver ≥18 years of age at the time of signing the informed consent; the study caregiver(s) must be able to recognize and observe the participant's seizures
* Participants with an established diagnosis of focal or generalized epilepsy or combined focal and generalized epilepsy with a documented history of stereotypical episodes of prolonged seizures that includes at least 1 of the following:

  1. Generalized seizure episodes starting with a flurry of absence seizures or myoclonic seizures with a minimum total duration of 5 minutes
  2. Episodes of a focal seizure with a minimum duration of 3 minutes
  3. Episodes of a focal seizure or a flurry of myoclonic seizures for at least 90 seconds followed by a generalized/bilateral tonic-clonic seizure with a minimum total duration of 3 minutes
* Prior to the Screening Visit, participant completed a study using Staccato alprazolam (such as EP0162 (NCT05077904), ENGAGE-E-001 (NCT03478982), or UP0100 (NCT04857307))

Exclusion Criteria:

* Participant has a current history of alcohol or drug use disorder, as defined in the Diagnostic and Statistical Manual of Mental Disorders 5, within the previous 1 year
* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) or comparable drugs (and/or an investigational device) as stated in this protocol or to albuterol (or similar bronchospasm rescue medication if needed to meet country-specific requirements)
* Participant has a history of convulsive (generalized tonic-clonic) status epilepticus in the 8 weeks prior to the Screening Visit
* Participant has a history or presence of known nonepileptic seizures which cannot be distinguished from qualifying epileptic seizures
* Participant has a clinically significant known airway hypersensitivity (eg, bronchospasm to known allergens, such as pollen, animals, or food) and/or acute respiratory signs/symptoms (eg, shortness of breath, wheezing on lung auscultation). NOTE: Participants with mild asthma who qualify for inclusion in the are allowed to be enrolled even though they have known airway hypersensitivity
* Participant has a clinically significant chronic pulmonary disorder other than mild asthma (eg, chronic obstructive pulmonary disease, restrictive lung diseases [including idiopathic pulmonary fibrosis]) and/or recent history or presence of hemoptysis or pneumothorax
* Participant has had a positive antigen test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and experienced moderate to severe signs/symptoms of respiratory distress necessitating hospitalization or outpatient treatment such as ambulatory oxygen, extensive treatment with inhaler medications, and/or oral medications for a duration of 4 weeks or more, unless full resolution occurred at least 6 months prior to Screening
* Participant has experienced a severe upper respiratory tract infection within 4 weeks or severe bronchitis/pneumonia within 3 months before the Screening Visit
* Participant has a history or presence of acute narrow-angle glaucoma
* Participant has a condition for which oral alprazolam is contraindicated as per the regional labeling
* Participant is taking any drug that is a strong CYP3A4 inhibitor, including azole antifungal agents (ketoconazole and itraconazole) and nefazodone
* Participant is taking any opioids or sedative hypnotics on a chronic basis
* Participant is taking nonselective beta blockers on a chronic basis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs) | From Baseline up to the End of Study Visit (up to 78 months)
  An Adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical product (IMP) and whether anticipated or unanticipated. A treatment-emergent adverse event (TEAE) is defined as any AE with a start date/time on or after the first IMP administration.
Frequency of TEAEs leading to withdrawal from study | From Baseline up to the End of Study Visit (up to 78 months)
  An Adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical product (IMP) and whether anticipated or unanticipated. A treatment-emergent adverse event (TEAE) is defined as any AE with a start date/time on or after the first IMP administration.
Frequency of serious TEAEs | From Baseline up to the End of Study Visit (up to 78 months)
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above

SECONDARY OUTCOMES:
Treatment success after investigational medicinal product (IMP) administration for seizures occurring within the first 12 months | From start of IMP treatment up to 12 months
  A responder after up to a maximum of 10 treated seizures will be defined as having a termination of seizure within 90 seconds after IMP dministration.
Treatment success after IMP administration with no recurrence after 2 hours for seizures during the first 12 months | From start of IMP treatment up to 12 months
  A responder after up to a maximum of 10 treated seizures will be defined as termination of seizure within 90 seconds after IMP administration and no recurrence of seizure(s) from IMP administration to 2 hours after IMP administration and no initiation of seizure rescue treatment from 90 seconds to 2 hours after IMP administration.
Frequency of respiratory TEAEs | From Baseline up to the End of Study Visit (up to 78 months)
  An Adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical product (IMP) and whether anticipated or unanticipated. A treatment-emergent adverse event (TEAE) is defined as any AE with a start date/time on or after the first IMP administration.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (143):
- United States (52):
  - Ep0165 50506, Phoenix, Arizona
  - Ep0165 50720, Scottsdale, Arizona
  - Ep0165 50494, Little Rock, Arkansas
  - Ep0165 50118, Downey, California
  - Ep0165 50416, La Jolla, California
  - Ep0165 50702, Long Beach, California
  - Ep0165 50722, Poway, California
  - Ep0165 50716, Sacramento, California
  - Ep0165 50367, New Haven, Connecticut
  - Ep0165 50088, Washington D.C., District of Columbia
  - Ep0165 50721, Boca Raton, Florida
  - Ep0165 50515, Gulf Breeze, Florida
  - Ep0165 50508, Jacksonville, Florida
  - Ep0165 50342, Jacksonville, Florida
  - Ep0165 50199, Miami, Florida
  - Ep0165 50676, Miami, Florida
  - Ep0165 50509, Orlando, Florida
  - Ep0165 50703, Rockledge, Florida
  - Ep0165 50308, Tampa, Florida
  - Ep0165 50323, Honolulu, Hawaii
  - Ep0165 50512, Boise, Idaho
  - Ep0165 50493, Chicago, Illinois
  - Ep0165 50375, Springfield, Illinois
  - Ep0165 50504, Fort Wayne, Indiana
  - Ep0165 50517, New Orleans, Louisiana
  - Ep0165 50615, Boston, Massachusetts
  - Ep0165 50047, Boston, Massachusetts
  - Ep0165 50507, St Louis, Missouri
  - Ep0165 50626, Neptune City, New Jersey
  - Ep0165 50299, New Brunswick, New Jersey
  - Ep0165 50497, Amherst, New York
  - Ep0165 50625, New Hyde Park, New York
  - Ep0165 50298, New York, New York
  - Ep0165 50490, New York, New York
  - Ep0165 50518, New York, New York
  - Ep0165 50034, Rochester, New York
  - Ep0165 50514, Charlotte, North Carolina
  - Ep0165 50715, Durham, North Carolina
  - Ep0165 50724, Portland, Oregon
  - Ep0165 50096, Philadelphia, Pennsylvania
  - Ep0165 50364, Philadelphia, Pennsylvania
  - Ep0165 50089, Philadelphia, Pennsylvania
  - Ep0165 50511, Pittsburgh, Pennsylvania
  - Ep0165 50491, Pittsburgh, Pennsylvania
  - Ep0165 50700, Chattanooga, Tennessee
  - Ep0165 50513, Memphis, Tennessee
  - Ep0165 50103, Nashville, Tennessee
  - Ep0165 50731, Austin, Texas
  - Ep0165 50714, Houston, Texas
  - Ep0165 50525, Houston, Texas
  - Ep0165 50473, Salt Lake City, Utah
  - Ep0165 50726, Winchester, Virginia
- Australia (3):
  - Ep0165 30016, Fitzroy
  - Ep0165 30030, Herston
  - Ep0165 30031, South Brisbane
- Bulgaria (5):
  - Ep0165 40650, Blagoevgrad
  - Ep0165 40708, Pazardzhik
  - Ep0165 40665, Pleven
  - Ep0165 40709, Pleven
  - Ep0165 40651, Sofia
- China (25):
  - Ep0165 20246, Beijing
  - Ep0165 20268, Beijing
  - Ep0165 20299, Beijing
  - Ep0165 20261, Changchun
  - Ep0165 20133, Chengdu
  - Ep0165 20137, Chengdu
  - Ep0165 20334, Chongqing
  - Ep0165 20179, Fuzhou
  - Ep0165 20124, Guangzhou
  - Ep0165 20264, Guangzhou
  - Ep0165 20269, Guangzhou
  - Ep0165 20300, Guangzhou
  - Ep0165 20022, Hangzhou
  - Ep0165 20320, Kunming
  - Ep0165 20258, Lanzhou
  - Ep0165 20267, Nanjing
  - Ep0165 20331, Nanning
  - Ep0165 20333, Qingdao
  - Ep0165 20292, Shanghai
  - Ep0165 20289, Shijiazhuang
  - Ep0165 20119, Suzhou
  - Ep0165 20257, Tianjin
  - Ep0165 20025, Wenzhou
  - Ep0165 20262, Zhanjiang
  - Ep0165 20251, Zhengzhou
- Czechia (5):
  - Ep0165 40670, Brno
  - Ep0165 40672, Ostrava - Poruba
  - Ep0165 40063, Prague
  - Ep0165 40671, Prague
  - Ep0165 40714, Prague
- Germany (7):
  - Ep0165 40683, Berlin
  - Ep0165 40685, Bielefeld
  - Ep0165 40023, Erlangen
  - Ep0165 40645, Frankfurt am Main
  - Ep0165 40689, Kehl
  - Ep0165 40529, Marburg
  - Ep0165 40724, München
- Hungary (4):
  - Ep0165 40666, Balassagyarmat
  - Ep0165 40673, Budapest
  - Ep0165 40704, Budapest
  - Ep0165 40653, Debrecen
- Italy (5):
  - Ep0165 40674, Genova
  - Ep0165 40144, Milan
  - Ep0165 40477, Pavia
  - Ep0165 40257, Roma
  - Ep0165 40675, Roma
- Japan (18):
  - Ep0165 20248, Fukuoka
  - Ep0165 20070, Hachioji-shi
  - Ep0165 20249, Hiroshima
  - Ep0165 20236, Hōfu
  - Ep0165 20239, Itami
  - Ep0165 20143, Kodaira
  - Ep0165 20315, Koshi-shi
  - Ep0165 20147, Kyoto
  - Ep0165 20243, Nagakute
  - Ep0165 20238, Niigata
  - Ep0165 20302, Osaka
  - Ep0165 20241, Ōmura
  - Ep0165 20316, Sapporo
  - Ep0165 20297, Shinjuku-ku
  - Ep0165 20240, Shizuoka
  - Ep0165 20242, Suita
  - Ep0165 20266, Tōon
  - Ep0165 20244, Yamagata
- Poland (7):
  - Ep0165 40707, Bydgoszcz
  - Ep0165 40677, Gdansk
  - Ep0165 40502, Krakow
  - Ep0165 40842, Krakow
  - Ep0165 40676, Lublin
  - Ep0165 40091, Nowa Sól
  - Ep0165 40678, Świdnik
- Spain (8):
  - Ep0165 40160, Barcelona
  - Ep0165 40157, L'Hospitalet de Llobregat
  - Ep0165 40540, Madrid
  - Ep0165 40352, Pamplona
  - Ep0165 40668, Seville
  - Ep0165 40453, Terrassa
  - Ep0165 40230, Valencia
  - Ep0165 40667, Valladolid
- United Kingdom (4):
  - Ep0165 40686, Birmingham
  - Ep0165 40735, Glasgow
  - Ep0165 40163, Oxford
  - Ep0165 40108, Salford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of reidentifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org